CLINICAL TRIAL: NCT06584812
Title: A Phase I Study to Evaluate the Pharmacokinetics, Pharmacodynamics and Safety in Healthy Subjects with Multiple Administration of Tiprogrel
Brief Title: Study to Assess Pharmacokinetics, Pharmacodynamics and Safety of Tiprogrel in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tianjin Institute of Pharmaceutical Research Co., Ltd (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: TY601A-P1-03
Record Dates: First submitted 2024-08-29; First posted 2024-09-05 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Acute Coronary Syndrome; Ischemic Stroke
MeSH Terms: conditions — Acute Coronary Syndrome; Ischemic Stroke | interventions — Clopidogrel; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tiprogrel-Clopidogrel-Ticagrelor (Other): Period 1: Dose 1 Tiprogrel; Period 2: Dose 2 Tiprogrel ; Period 3: Clopidogrel; Period 4: Ticagrelor
  Interventions: Drug: Tiprogrel; Drug: Clopidogrel; Drug: Ticagrelor

INTERVENTIONS:
Drug: Tiprogrel — Period 1: Dose 1 Tiprogrel, loading dose of Tiprogrel followed by daily maintenance dose until Day 8.
Drug: Tiprogrel — Period 2: Dose 2 Tiprogrel ; loading dose of Tiprogrel followed by daily maintenance dose until Day 8.
Drug: Clopidogrel — Period 3: Clopidogrel; loading dose of Clopidogrel followed by daily maintenance dose until Day 8.
Drug: Ticagrelor — Period 4: Ticagrelor; loading dose of Ticagrelor followed by daily maintenance dose until Day 8.

SUMMARY:
This study is designed to evaluate the pharmacokinetics, pharmacodynamics and safety in healthy subjects with multiple administration of Tiprogrel.

DETAILED DESCRIPTION:
Tiprogrel is a novel oral P2Y12 receptor antagonist.This study is to evaluate the pharmacokinetics, pharmacodynamics and safety in healthy subjects with multiple administration of Tiprogrel, and compare pharmacokinetics /pharmacodynamic of Tiprogrel,Clopidogrel and Ticagrelor.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female Healthy Subjects
2. Subject has the ability and willingness to comply with study procedures and follow-up examination.

3：18 to 50 years of age (including the threshold) 4: Body mass index (BMI) ≥ 19.0 to ≤ 28.0 kg/m2; total body weight of male subject ≥ 50 kg at Screening; total body weight of female subject ≥ 45 kg at Screening; 5：Medically healthy based on their medical history, and physical examination, clinical laboratory test results, ECGs, and vital sign measurements as determined by the Investigator at Screening; 6: Female subjects are not pregnant or breastfeeding, and the fertile female and male subjects must agree to follow instructions for method(s) of contraception.

Exclusion Criteria:

1. History or presence of metabolic, allergy, dermatology, liver, kidney, hematology, cardiovascular, gastrointestinal, nervous, respiratory, endocrine or psychiatric diseases.
2. History or presence of obviously active bleeding, or coagulation or bleeding disorders, or any skin petechiae, or thrombus, or spontaneous bleeding.
3. Subject with history of allergy to a variety of drugs, or has a known or suspected hypersensitivity to tiprogrel or other anti-platelet drugs
4. Subjects who had a history of major surgery within 3 months before the trial or planned to undergo surgery during the study period.
5. Subjects who have lost or donated ≥ 400 mL blood or received blood transfusion or used blood products within three months, or subjects with clinically significant anemia based on the judgment of the Investigator
6. Subjects with systolic blood pressure of > 140 mmHg or < 90 mmHg, diastolic blood pressure of > 90 mmHg or < 60 mmHg
7. Subjects with 12-lead ECG examination: QTcF > 450 msec
8. Platelet count (PLT) value, beyond the laboratory's reference range
9. Activated partial thromboplastin time (APTT) and Prothrombin Time (PT), beyond the laboratory's reference range
10. ALT, AST, γ-GGT, ALP and TBIL value >1.5 times the upper limit of normal value
11. Subjects with positive results at screening for HIV, syphilis, HBsAg, or HCV
12. Subjects who have taken aspirin/other nonsteroidal anti-inflammatory drugs (NSAIDs) or other drugs that may affect coagulation function within 2 weeks before the trial
13. Subjects who have taken prescription drugs/products or herbs within 2 weeks or 5 half-lives (whichever is longer) before the trial;or taken OTC drugs/products within 7 days before the trial.
14. Subjects who have received live or attenuated vaccines within 1 month prior to receiving the study drug or expected to receive vaccines during the study period
15. Subjects who have ingested investigational drug within 3 months or 5 half-lives prior to the first study drug dose
16. Subjects who have participated in another clinical trial within 3 months or 5 half-lives prior to the first study drug dose;
17. Consumption of any known liver enzyme inducers/inhibitors within 30 days prior to the first study drug dose;
18. Have a history of drug addiction or drug abuse within 1 year prior to screening;
19. Positive results for alcohol, or cotinine, or urine for drugs test in screening or admission;
20. Subject with alcohol consumption defined as > 21 units per week for men and > 14 units per week for woman;
21. Use of tobacco or nicotine-containing products within 1 month prior to screening;
22. CYP2C19 poor metabolizer;
23. Subjects with a history of fainting needle or blood;
24. Subjects who are not suitable to participate in this experiment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
PK parameters： Cmax | Day 1 to Day 9 in each period
  Maximum Concentration of Tiprogrel 's active metabolite
PK parameters： Cmax | Day 1 to Day 9 in each period
  Maximum Concentration of Clopidogrel 's active metabolite
PK parameters： AUC | Day 1 to Day 9 in each period
  Area under the plasma concentration curve of Tiprogrel 's active metabolite
PK parameters： AUC | Day 1 to Day 9 in each period
  Area under the plasma concentration curve of Clopidogrel 's active metabolite
PK parameters： Tmax | Day 1 to Day 9 in each period
  Time to maximum concentration of Tiprogrel 's active metabolite
PK parameters： Tmax | Day 1 to Day 9 in each period
  Time to maximum concentration of Clopidogrel 's active metabolite
PK parameters： T1/2 | Day 1 to Day 9 in each period
  Half life of Tiprogrel 's active metabolite
PK parameters： T1/2 | Day 1 to Day 9 in each period
  Half life of Clopidogrel 's active metabolite
PD parameters: Adenosine Diphosphate(ADP)-induced P2Y12 Receptor-mediated platelet aggregation of Tiprogrel | Day 1 to Day 14 in each period
  ADP-induced platelet reaction unit represents the rate and extent of ADP-stimulated platelet aggregation
PD parameters: Adenosine Diphosphate(ADP)-induced P2Y12 Receptor-mediated platelet aggregation of Clopidogrel | Day 1 to Day 14 in each period
  ADP-induced platelet reaction unit represents the rate and extent of ADP-stimulated platelet aggregation
PD parameters: Adenosine Diphosphate(ADP)-induced P2Y12 Receptor-mediated platelet aggregation of Ticagrelor | Day 1 to Day 14 in each period
  ADP-induced platelet reaction unit represents the rate and extent of ADP-stimulated platelet aggregation
Safety parameters: Number of Participants With Treatment-Related Adverse Events | Day 1 to Day 14 in each period

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hosptial, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No